CLINICAL TRIAL: NCT00808795
Title: Efficacy of N-Acetylcysteine in Prevention of Contrast-Induced Nephropathy After Cardiac Catheterization in Patients With Diabetes Mellitus and Chronic Kidney Disease: A Randomized Clinical Trial
Brief Title: Efficacy of N-Acetylcysteine in Prevention of Post-Catheterization Contrast-Induced Nephropathy in Diabetic Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Tehran University of Medical Sciences, Nephrology Department of Dr. Shariati Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 487
Record Dates: First submitted 2008-12-13; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Radiocontrast-Induced Nephropathy; Chronic Kidney Disease; Diabetes Mellitus
Keywords: Acute kidney injury; contrast-induced nephropathy; Chronic kidney disease; Diabetes mellitus; N-acetylcysteine
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Acute Kidney Injury | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (Experimental)
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — NAC is to be orally administered at the dose of 600mg twice a day, starting 24h before the procedure (two doses before and two doses after the procedure).
  Arms: N-acetylcysteine
Drug: Placebo — Placebo of NAC is to be orally administered at the dose of 600mg twice a day, starting 24h before the procedure (two doses before and two doses after the procedure).
  Arms: Placebo

SUMMARY:
* Contrast-induced nephropathy (CIN) is the third most common cause of hospital acquired acute kidney injury, accounting for 10% of all cases.
* The pathophysiology of CIN is unclear. Possible mechanisms involve

  1. Renal tubular injury by oxygen free radicals
  2. Reducing renal blood flow which leads to acute tubular necrosis. Since N-acetylcysteine is an antioxidant as well as a vasodilator, it may work in two distinct ways, by preventing reduction in renal blood flow or contrast-induced oxidative damage.
* The purpose of this study is to evaluate the efficacy of N-acetylcysteine compared to placebo for the contrast-induced nephropathy prevention.

DETAILED DESCRIPTION:
* Contrast-induced nephropathy (CIN) is the third most common cause of hospital acquired acute kidney injury, accounting for 10% of all cases. Nevertheless, use of radiocontrast media has been associated with increased in-hospital morbidity, mortality, and costs of medical care, long admission, especially in patients needing dialysis. With the increasing use of contrast media in diagnostic and interventional procedures, it has become one of the major challenges encountered during routine cardiovascular practice.
* Patients at the greatest risk for CIN can be defined as those have preexisting impaired renal function and diabetes mellitus with incidence estimated to be as high as 50%. Preventive therapies primarily include limitation of contrast exposure, intravenous volume expansion with a saline solution, and use of a low- or iso-osmolality contrast media.
* However, since these measures provide incomplete protection for CIN, interest has emerged in a number of adjunction short-term pharmacotherapy methods. Among them, N-acetylcysteine (NAC) has been of considerable interest. Up to now, several clinical studies and meta-analysis have been performed to assess the efficacy of NAC in prevention of CIN.
* In spite of heterogeneity regarding efficacy of administration of NAC, several studies have advised the use of NAC, especially in high risk patients, with regard to its low cost, availability and few side effects. Since administration of NAC necessitates earlier and longer admission of patients, particularly in intravenous use, it can increase the health care costs. In addition, there are evidences that this intervention can even be harmful in patients with diabetes mellitus.
* So, it seems that we need more evidences about the efficacy and cost-effectiveness of NAC in patients at high risk for development of CIN to make rational clinical decisions for individual patients as well as policy decisions for the health of the general public.

ELIGIBILITY:
Inclusion Criteria:

Patients who have all of the following criteria:

* Aged older than 18 years old
* A history of diabetes mellitus for at least one year
* chronic kidney disease, defined as serum creatinine concentration >=1.5mg/dL for men and >=1.4mg/dL for women.

Exclusion Criteria:

* Acute coronary syndrome requiring primary or rescue coronary intervention within less than 12h
* Cardiogenic shock
* Current peritoneal or hemo-dialysis
* A known allergy to NAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Incidence of CIN, defined as increase in serum creatinine concentration>=0.5mg/dL(44.2micromol/L) or >=25% above baseline. | 48 hours after exposure to contrast medium

SECONDARY OUTCOMES:
Change in serum creatinine | 48 hours after exposure to contrast medium
Change in serum urea nitrogen | 48 hours after exposure to contrast medium
Change in Glomerular filtration rate(GFR) | 48 hours after exposure to contrast medium

CONTACTS AND LOCATIONS:
Overall Officials: Manouchehr - Amini, MD, Study Director — Tehran University of Medical Sciences, Nephrology Department of Dr. Shariati Hospital
Locations (1):
- Tehran Heart center, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Amini M, Salarifar M, Amirbaigloo A, Masoudkabir F, Esfahani F. N-acetylcysteine does not prevent contrast-induced nephropathy after cardiac catheterization in patients with diabetes mellitus and chronic kidney disease: a randomized clinical trial. Trials. 2009 Jun 29;10:45. doi: 10.1186/1745-6215-10-45. PMID 19563648